CLINICAL TRIAL: NCT04720235
Title: A Follow On Community Testing Study To Evaluate The Performance of the Lucira COVID-19 All-In-One Test Kit As Compared To The Hologic Panther Fusion SARS-CoV-2 RT-PCR Assay Among Asymptomatic Subjects
Brief Title: A Follow On Community Testing Study To Evaluate The Performance of the Lucira COVID-19 All-In-One Test Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucira Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07A-CLI-007
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subject Self-Collection and Specimen Testing (Other): Subjects will be provided with the Lucira COVID-19 Test Kit and collect one (1) nasal swab according to the QRI and test the sample on the Lucira COVID-19 All-In-One Test. HCP will observe subject during this process and document any observations and deviations from the QRI.
  Interventions: Device: Lucira COVID-19 All-In-One test kit

INTERVENTIONS:
Device: Lucira COVID-19 All-In-One test kit — The Lucira COVID-19 All-In-One Test Kit is intended to detect the novel coronavirus SARS-CoV-2 that causes COVID-19 in nasal swab samples. This test is a single-use test kit that determines whether there is active shedding of the virus which causes COVID-19. This test utilizes a molecular amplification technology for the detection of SARS-CoV-2 RNA.
  Positive results are indicative of active infection with SARS-CoV-2. Persons who test positive should self-isolate and seek care from their healthcare provider.
  Negative results do not preclude SARS-CoV-2 infection. Persons who continue to experience COVID-like symptoms should seek follow up care from their healthcare provider

SUMMARY:
To evaluate the performance of the FDA EUA authorized Lucira COVID-19 All-In-One Test Kit for the qualitative detection of SARS-CoV-2 virus in nasal swab samples as compared to a known high sensitivity EUA RT-PCR among asymptomatic individuals. The comparator assay for this study is the Hologic Panther Fusion SARS-CoV-2 RT-PCR Assay.

DETAILED DESCRIPTION:
This Lucira COVID-19 All-In-One Test Kit recently received FDA Emergency Use Authorization (EUA) for prescription home use with self-collected nasal swab samples in individuals aged 14 and older who are suspected of COVID-19 by their healthcare provider. The basis for this FDA EUA authorization was Lucira Health's first Community Testing study (07A-CLI-006) conducted among individuals suspected of COVID-19. This follow on performance study will be used to establish the performance of the Lucira COVID-19 All-In-One Test Kit as compared to a known high sensitivity RT-PCR molecular assay among asymptomatic individuals. The results of this study will be used to support an expanded indication for the Lucira COVID-19 All-In-One Test Kit among asymptomatic individuals.

This performance study will include the collection of subject demographics and nasal swabs self-collected by study subjects at community-based locations with trained medical staff oversight.

After determining subject eligibility and following the completion of the informed consent process, each subject will receive a unique study identification number.

A subject's participation in this study will consist of one study visit with one collection event. The subject self-collects a nasal swab sample and runs the Lucira COVID-19 All-In-One Test Kit according to the FDA EUA authorized package insert instructions.

Subject will be observed during the swabbing collection by the study staff and study staff will document collection details and any collection issues. Nasal swabs obtained from self-collection will be discarded after having been used for testing per the instructions. Study staff will interpret and share the Lucira COVID-19 All-In-One Test Kit result with study subjects.

Following the Lucira COVID-19 All-In-One Test Kit self-collection will be an additional swab collection for reference method testing. One (1) additional NS specimen will be self-collected, prepared in Transport Medium and sent to the reference laboratory as directed by the Study Operations Manual.

Each collection may have a maximum of two swabs, including retests, for a maximum of four swabs per visit.

ELIGIBILITY:
Inclusion Criteria

1. Ages 14-75
2. Must be able to read and write in English
3. Must be willing to try rapid COVID-19 test and self-collect a nasal swab sample in both nostrils

Exclusion Criteria

* Currently suffering from nasal trauma such as a nosebleed
* Received a nasal rinse/wash/aspirates in past 12 hours
* Currently experiencing any of the CDC COVID-19 symptoms:

  * Fever
  * Cough
  * Shortness of breath or difficulty breathing
  * Fatigue
  * New loss of taste or smell
  * Muscle or body aches
  * Headache
  * Sore throat
  * Congestion or runny nose
  * Nausea or vomiting
  * Diarrhea

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 Prevalence Rate / Expected Values counts | 3 months
  Study prevalence of SARS-CoV-2 will be summarized by counts and grouped by age
COVID-19 Prevalence Rate / Expected Values percentages | 3 Months
  Study prevalence of SARS-CoV-2 will be summarized by percentages and grouped by age

SECONDARY OUTCOMES:
Collection Performance/ Incidence Rate counts | 3 Months
  Study observations will be summarized by counts:
  * Self-Collection, Self-tested
  * User Experience
Collection Performance/ Incidence Rate percentages | 3 Months
  Study observations will be summarized by percentages:
  * Self-Collection, Self-tested
  * User Experience
Sensitivity and specificity | 3 Months
  Sensitivity and specificity along with their associated 2-sided Wilson Score 95% Confidence Intervals will be estimated for SARS-CoV-2, on the Lucira COVID-19 All-In-One Test in comparison to the reference test

OTHER OUTCOMES:
Invalid Rate | 3 Months
  The invalid rates, along with their associated 2-sided Wilson Score 95% Confidence Intervals will be estimated for SARS-CoV-2 on the Lucira COVID-19 All-In-One Test

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Kochhar, MD, Principal Investigator — Neeraj Kochhar Family Medicine
Locations (1):
- Neeraj Kochhar Family Medicine, Los Gatos, California, United States

IPD SHARING:
Plan to Share IPD: No